CLINICAL TRIAL: NCT01290900
Title: A Single-centre, Randomised, Double-blind, Placebo-controlled, Four Way Crossover Phase I Study to Investigate the Effect on QT/QTc Interval of a Single Dose of Intravenous Ceftazidime NXL104 (3000/2000 mg) or Ceftaroline Fosamil NXL104 (1500/2000 mg), Compared With Placebo, Using Open-label Moxifloxacin (Avelox®) as a Positive Control, in Healthy Male Volunteers
Brief Title: A Single-centre, Randomised, Double-blind, Placebo-controlled, Four Way Crossover Phase I Study to Investigate the Effect on QT/QTc Interval of Ceftazidime NXL104 or Ceftaroline Fosamil NXL104, Compared With Placebo, Using Moxifloxacin (Avelox®) as a Positive Control, in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Paul Newell / Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D4280C00007
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Healthy Male Volunteers
Keywords: NXL104; CAZ104; Ceftazidime; CXL104; Ceftaroline; Healthy Male Volunteers; Phase 1; OT; Single Dose Study
MeSH Terms: interventions — avibactam; Ceftaroline; Ceftazidime; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CXL104 (Experimental): 2000 mg NXL104 + 1500 mg Ceftaroline (IV)
  Interventions: Drug: NXL104; Drug: Ceftaroline
- CAZ104 (Experimental): Placebo Infusion (saline) + 2000 mg NXL104 + 3000 mg Ceftazidime (IV)
  Interventions: Drug: NXL104; Drug: Placebo Infusion; Drug: Ceftazidime
- Moxifloxacin (Active Comparator): Moxifloxacin 400mg (1 tablet)
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator): Placebo Infusion (saline)
  Interventions: Drug: Placebo Infusion

INTERVENTIONS:
Drug: NXL104 — IV Solution
  Arms: CAZ104; CXL104
Drug: Ceftaroline — IV Solution
  Arms: CXL104
Drug: Placebo Infusion — IV Saline
  Arms: CAZ104; Placebo
Drug: Ceftazidime — IV Solution
  Arms: CAZ104
Drug: Moxifloxacin — Tablet (1)
  Arms: Moxifloxacin

SUMMARY:
This is a single dose study in healthy male volunteers to investigate the effect of high doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent prior to any study specific procedures
* Healthy male volunteers aged 18 to 45 years (inclusive) with suitable veins for cannulation or repeated venepuncture
* Have a body mass index (BMI) between 19 and 30 kg/m2 and a body weight between 60 and 100 kg
* Be a non-smoker or ex-smoker who has stopped smoking (or using other nicotine products) for more than 3 months prior to the start of the study

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
* Any clinically significant abnormalities in physical examination, clinical chemistry, haematology or urinalysis results as judged by the Investigator
* Abnormal vital signs, after 10 minutes supine rest, defined as any of the following: Systolic blood pressure (SBP) greater than 140 mmHg, Diastolic blood pressure (DBP) greater than 90 mmHg, Heart rate less than 40 or greater than 85 beats per minute - at Visit 1
* Prolonged QTcF >450 ms or shortened QTcF <340 ms
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes. This includes volunteers with any of the following: Clinically significant PR (PQ) interval prolongation, Intermittent second or third degree AV block (Mobitz II type 1, Wenchebach during sleep is not disqualifying), Incomplete, full or intermittent bundle branch block (QRS less than 110 ms with normal QRS and T wave morphology is acceptable if there is no evidence of left ventricular hypertrophy), Abnormal T wave morphology, particularly in the protocol defined primary lead

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of supratherapeutic doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval (QTcF). | 12-lead dECG will be performed pre-dose
To investigate the effect of supratherapeutic doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval (QTcF). | 12-lead dECG at 30 min after starting dosing.
To investigate the effect of supratherapeutic doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval (QTcF). | 12-lead dECG at 60 min after starting dosing.
To investigate the effect of supratherapeutic doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval (QTcF). | 12-lead dECG at 90 min after starting dosing.
To investigate the effect of supratherapeutic doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval (QTcF). | 12-lead dECG at 2 hour after starting dosing.
To investigate the effect of supratherapeutic doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval (QTcF). | 12-lead dECG at 3 hour after starting dosing.
To investigate the effect of supratherapeutic doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval (QTcF). | 12-lead dECG at 4 hour after starting dosing.
To investigate the effect of supratherapeutic doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval (QTcF). | 12-lead dECG at 6 hour after starting dosing.
To investigate the effect of supratherapeutic doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval (QTcF). | 12-lead dECG at 8 hour after starting dosing.
To investigate the effect of supratherapeutic doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval (QTcF). | 12-lead dECG at 12 hour after starting dosing.
To investigate the effect of supratherapeutic doses of ceftazidime NXL104 (CAZ104) or ceftaroline fosamil NXL104 (CXL104) on the QT interval (QTcF). | 12-lead dECG at 24 hour after starting dosing.

SECONDARY OUTCOMES:
To investigate the effect of CAZ104 and CXL104, on additional ECG variables (heart rate, RR, PR, QRS, QT, and QTcB). | 12-lead dECG will be performed pre-dose
To investigate the effect of CAZ104 and CXL104, on additional ECG variables (heart rate, RR, PR, QRS, QT, and QTcB). | 12-lead dECG at 30 min after starting dosing.
To investigate the effect of CAZ104 and CXL104, on additional ECG variables (heart rate, RR, PR, QRS, QT, and QTcB). | 12-lead dECG at 60 min after starting dosing.
To investigate the effect of CAZ104 and CXL104, on additional ECG variables (heart rate, RR, PR, QRS, QT, and QTcB). | 12-lead dECG at 90 min after starting dosing.
To investigate the effect of CAZ104 and CXL104, on additional ECG variables (heart rate, RR, PR, QRS, QT, and QTcB). | 12-lead dECG at 2 hour after starting dosing.
To investigate the effect of CAZ104 and CXL104, on additional ECG variables (heart rate, RR, PR, QRS, QT, and QTcB). | 12-lead dECG at 3 hour after starting dosing.
To investigate the effect of CAZ104 and CXL104, on additional ECG variables (heart rate, RR, PR, QRS, QT, and QTcB). | 12-lead dECG at 4 hour after starting dosing.
To investigate the effect of CAZ104 and CXL104, on additional ECG variables (heart rate, RR, PR, QRS, QT, and QTcB). | 12-lead dECG at 6 hour after starting dosing.
To investigate the effect of CAZ104 and CXL104, on additional ECG variables (heart rate, RR, PR, QRS, QT, and QTcB). | 12-lead dECG at 8 hour after starting dosing.
To investigate the effect of CAZ104 and CXL104, on additional ECG variables (heart rate, RR, PR, QRS, QT, and QTcB). | 12-lead dECG at 12 hour after starting dosing.
To investigate the effect of CAZ104 and CXL104, on additional ECG variables (heart rate, RR, PR, QRS, QT, and QTcB). | 12-lead dECG at 24 hour after starting dosing.
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken pre-dose
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 30 min after starting dosing
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 60 min after starting dosing
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 75 min after starting dosing
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 90 min after starting dosing
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 2 hour after starting dosing
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 3 hour after starting dosing
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 4 hour after starting dosing
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 6 hour after starting dosing
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 8 hour after starting dosing
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 12 hour after starting dosing
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 18 hour after starting dosing
To assess the PK of NXL104, ceftaroline, ceftazidime and moxifloxacin by determination where applicable of Cmax, tmax, AUC(0-t), AUC, t½, CL, CL/F, Vss, and Vz/F. | Blood samples will be taken at 24 hour after starting dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newell, MD, Study Director — AstraZeneca; David Mathews, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Das S, Armstrong J, Mathews D, Li J, Edeki T. Randomized, placebo-controlled study to assess the impact on QT/QTc interval of supratherapeutic doses of ceftazidime-avibactam or ceftaroline fosamil-avibactam. J Clin Pharmacol. 2014 Mar;54(3):331-40. doi: 10.1002/jcph.199. Epub 2013 Oct 22. PMID 24150927